CLINICAL TRIAL: NCT03295435
Title: Associations Between the Composition of Functional Tooth Units and Nutrient Intake in Older Men: the Concord Health and Ageing in Men Project.
Brief Title: Composition of Functional Tooth Units and Nutrient Intake in Older Men
Acronym: CHAMP
Status: Completed | Type: Observational
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Other Study IDs: 301916
Record Dates: First submitted 2017-09-24; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Oral Health of Older Men; Dietary Assessment of Older Men
Keywords: Diet; Oral Health; Nutrition; Dentition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Composition of functional tooth units — Composition of functional tooth units measured by trained oral health therapists and was categorised into 3 groups:
  Group A: Natural units only Group B: Natural & Prosthetic units present Group C: No natural units present

SUMMARY:
Various definitions of poor dentition in older adults has been linked with inadequate intake of nutrients and poor diet quality. This study aims to look at the associations between poor dentition as defined by the composition of functional tooth units, and dietary intake of nutrients in community dwelling older men.

DETAILED DESCRIPTION:
Poor dentition, defined by numbers of teeth, functional tooth units or edentulism has been previously shown to be associated with poor intakes of nutrients in older adults, including but not limited to vitamin C, calcium, fibre, protein, zinc and folate. Similar findings have been found when poor dentition is defined by the presence of a prosthesis. Reasons for this inverse relationship include poor denture quality, reduced chewing capacity, or the inadequacy of prosthesis to replace natural teeth.

However limited studies have looked at how the composition (natural verses prosthetic) of functional tooth units is associated with nutrient intake. A cross sectional analysis of a cohort of male older adults, participating in an ongoing longitudinal study, was conducted to investigate nutrition and oral health associations, including the relationship between the composition of functional tooth units and nutrient intake.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Moved inter or intrastate (moved out of study area)
* Death
* Refused to participate
* previously withdrawn

Min Age: 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population is a subset of a ongoing longitudinal study, that start in 2005. Men over the age of 70 years on the electoral roll for geographical locations within the Canada Bay area of Sydney, NSW were invited to participate. The only exclusion criteria was living in an aged care facility at time of recruitment.
  The follow up this study is based on, invited participants to be involved in a fourth wave of assessments. Anyone who had moved into an aged care facility was included. However those who had moved outside of the Sydney, had died, previously withdrawn or refused to participate, (but remained active), were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2016-07-13 (Actual); Study Completion 2016-07-13 (Actual)

PRIMARY OUTCOMES:
Dietary intake of nutrients | 45 minute interview on 1 day (cross-sectional).
  A diet history was performed, and data entered into a database which provided daily average nutrient intakes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Cumming, PhD, Principal Investigator — University of Sydney
Locations (1):
- The Centre for Education and Research on Ageing, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data is be available for researchers.
Time Frame: Data is currently available
Access Criteria: Data access request will be reviewed by Chief Investigators. All requester's will be required to sign a data access agreement.

REFERENCES:
- [Background] de Andrade FB, de Franca Caldas A Jr, Kitoko PM. Relationship between oral health, nutrient intake and nutritional status in a sample of Brazilian elderly people. Gerodontology. 2009 Mar;26(1):40-5. doi: 10.1111/j.1741-2358.2008.00220.x. Epub 2008 Feb 19. PMID 18298586
- [Background] Hildebrandt GH, Dominguez BL, Schork MA, Loesche WJ. Functional units, chewing, swallowing, and food avoidance among the elderly. J Prosthet Dent. 1997 Jun;77(6):588-95. doi: 10.1016/s0022-3913(97)70100-8. PMID 9185051
- [Background] Ervin RB, Dye BA. The effect of functional dentition on Healthy Eating Index scores and nutrient intakes in a nationally representative sample of older adults. J Public Health Dent. 2009 Fall;69(4):207-16. doi: 10.1111/j.1752-7325.2009.00124.x. PMID 19453869
- [Background] Shinkai RS, Hatch JP, Rugh JD, Sakai S, Mobley CC, Saunders MJ. Dietary intake in edentulous subjects with good and poor quality complete dentures. J Prosthet Dent. 2002 May;87(5):490-8. doi: 10.1067/mpr.2002.124093. PMID 12070511
- [Background] Ueno M, Yanagisawa T, Shinada K, Ohara S, Kawaguchi Y. Masticatory ability and functional tooth units in Japanese adults. J Oral Rehabil. 2008 May;35(5):337-44. doi: 10.1111/j.1365-2842.2008.01847.x. PMID 18405269